CLINICAL TRIAL: NCT04047407
Title: Pain Response Characteristics to Different Doses of Suprathreshold Pressure Stimulation in Fibromyalgia Subjects
Brief Title: Suprathreshold Pressure Pain Stimulation in Fibromyalgia
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Other Study IDs: Suprathresholds fibromyalgia
Record Dates: First submitted 2019-07-30; First posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Fibromyalgia
Keywords: Reffered pain; Pain sensitivity; Fibromyalgia; Suprathreshold; Central sensitization
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibromyalgia
  Interventions: Device: Suprathreshold pain stimulation
- Healthy volunteers
  Interventions: Device: Suprathreshold pain stimulation

INTERVENTIONS:
Device: Suprathreshold pain stimulation — Suprathreshold pain stimulation will be applied in the infraspinatus muscle (point equidistant between the midpoint of the spine of the scapula, the inferior angle of the scapula and the midpoint of the medial border of the scapula) with a pressure algometer (Force Ten ™, Wagner Instruments, USA). Four suprathreshold pressure stimulations (pressure pain threshold + 20%, +30%, +40% and +50%) will be made for 60 seconds, with a minimum rest of 5 minutes between each stimulation.
  The sequence of stimulation (ascending or descending) will be randomized.

SUMMARY:
The purpose of this study is to investigate the induced-pain characteristics after suprathreshold pressure stimulation at different intensities in fibromyalgia subjects, compared with healthy volunteers.

DETAILED DESCRIPTION:
Fibromyalgia syndrome is a chronic painful, non-inflammatory rheumatic disease with a high negative impact on the quality of life, and is characterized by widespread pain, fatigue and generalised hyperalgesia on examination, symptoms that can be the consequence of central sensitization.

Despite several methods have successfully addressed this increased responsiveness of nociceptive neurons in the central nervous system, there is a lack of consensus about how to systematically perform them and those that are more appropriated for different syndromes. Therefore, investigating appropriate simple methods to assess clinical manifestations of central sensitization is relevant in the assessment of fibromyalgia.

The present study aims to investigate the pain response after suprathreshols pressure stimulation in fibromyalgia subjects compared with healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Fullfilled the American Collegue of Rheumathology criteria for fibromyalgia.
* Understanding of spoken and written Spanish.

Exclusion Criteria:

* Diagnosed psychiatric pathology.
* Rheumatic pathology not medically controlled.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subject recruitment will be carried out in a local fibromyalgia association. Healthy volunteers will be recruitment among hospital and university workers.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-09-18 (Estimated); Study Completion 2019-09-18 (Estimated)

PRIMARY OUTCOMES:
Referred pain induced area after suprathreshold pressure stimulation | Inmediately after each stimulation
  After each stimulation (120%, 130%, 140% and 150%), the subject should draw the induced pain area on a digital bodychart using the Navigate Pain application (Navigate Pain, Aalborg University, Denmark). The size of the areas of referred pain will be extracted in pixels.

SECONDARY OUTCOMES:
Pain intensity | Inmediately after each stimulation
  It will be measured with a visual analog scale (VAS) of 100 millimeters in length. The subject has to indicate the level of pain he feels, being 0 the absence of pain and 100 the maximum imaginable.
Body regions afected by pain after suprathreshold pressure stimulation | Inmediately after each stimulation
  The digital body chart will be divided into 15 different regions: (1) posterior head and neck area; (2) supraspinal area; (3) infraspinatus area; (4) posterior shoulder area; (5) back area; (6) posterior arm area; (7) posterior forearm area; (8) posterior hand area; (9) anterior head and neck area; (10) supraclavicular area; (11) chest area; (12) anterior shoulder area; (13) anterior arm area; (14) anterior forearm area; (15) anterior hand area. The total number of body regions afected by pain will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Arroyo Fernández, MsC, PT, Principal Investigator — University of Castilla-La Mancha
Locations (1):
- Hospital General Nuestra Señora del Prado, Talavera de la Reina, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No